CLINICAL TRIAL: NCT05462808
Title: ART Restorations With High-viscosity Glass-ionomer Cement Versus Hall Technique in Primary Molars
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esra Oz (Other)
Responsible Party: Sponsor-Investigator, Esra Oz, Pediatric department, Suleyman Demirel University
Organization: Suleyman Demirel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/157
Record Dates: First submitted 2022-07-04; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Primary Teeth Retained

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atraumatic Restorative Treatment restorations with high-viscosity glass ionomer cement (Experimental): Under cotton roll isolation, teeth were restored with EQUIA Forte cement. A layer of EQUIA Forte Coat was applied with a microbrush on surface and then light cured for 20 s
  Interventions: Drug: High viscosity glass ionomer cement
- restorations with Hall technique (Experimental): In the Hall technique group, the deposits on the occlusal surface of the teeth were gently removed, SSC (3M ESPE, St. Paul, USA) was placed and were cemented using GIC. The crown was pressed tightly.
  Interventions: Device: Stainless steel crown

INTERVENTIONS:
Drug: High viscosity glass ionomer cement — High viscosity glass ionomer cement
  Other Names: EQUIA Forte (GC Corp., Leuven, BE)
  Arms: Atraumatic Restorative Treatment restorations with high-viscosity glass ionomer cement
Device: Stainless steel crown — Stainless steel crown
  Other Names: 3M ESPE, St. Paul, USA
  Arms: restorations with Hall technique

SUMMARY:
Primary molars are the teeth with the highest caries tendency among primary teeth due to their anatomical features such as wide and flat interface areas. However, some difficulties are encountered during the removal of caries due to the structural features of primary molars and the young age of the child. Therefore, in the treatment of primary molars, Atraumatic Restorative Treatment (ART), in which the soft parts of the carious lesion are cleaned with the help of a sharp hand tool and restored with an adhesive glass ionomer cement (GIC) that releases fluoride, in the following years, the deciduous teeth were removed with a minimally invasive approach. Hall technique, in which a stainless steel crown (SSC) is placed without preparation for treatment, has come to the fore.

DETAILED DESCRIPTION:
Many restorative materials, especially GIC, have been used for ART procedures, and with the advancing technology, high-viscosity glass ionomer cements with improved mechanical and chemical properties have emerged. In recent years, zinc-added HVGICs and nano-filled resin-modified HVGICs have been introduced.

The Hall Technique has been suggested in the treatment of asymptomatic decayed primary molars in anxious and fearful patients to ensure patient cooperation. In this technique, it is aimed to stop the progression of caries by covering the carious deciduous molars with SSC and cutting their relationship with the oral environment, without the need for local anesthesia and tooth preparation. Thus, as the bacteria cannot use the carbohydrates in the oral environment, the number of bacteria in the environment will also decrease.

ELIGIBILITY:
Inclusion Criteria:

* children with no systemic disease,
* children who had a Frankl Behavioral Scale score 2,
* children who have no occlusal problems or bad habits,
* children presenting between 2-5 caries lesion in primary molars.

Exclusion Criteria:

* teeth with presence of radyolusens in furcation and/or periradicular areas,
* teeth with pathologic resorption and internal/external resorption

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Hall technique | up to 18 months
  The restorations were scored as Alpha (A), clinically ideal restoration ''successful''; Bravo (B), clinically ''acceptable''; Charlie (C), clinically unacceptable restoration ''unsuccessful''. Outcomes criteria for assessment of the Hall Technique were made according to Innes et al.

SECONDARY OUTCOMES:
Atraumatic restorative treatment | up to 18 months
  Clinical evaluations of teeth treated with ART using EQUIA Forte were performed according to the modified USPHS criteria established by a modification of the United States Public Health Service (USPHS) clinical evaluation criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Oz, Study Director — Suleyman Demirel University Pediatric Dentistry
Locations (1):
- Suleyman Demirel University Faculty of Dentistry Pediatric Dentistry Department, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No